CLINICAL TRIAL: NCT07126574
Title: Research Protocol for Evaluating the Diagnostic Utility of SAA, Procalcitonin, Presepsin, CRP, and Routine Blood Biomarkers in Adult Burn Patients With Sepsis in the Intensive Care Unit
Brief Title: Evaluating the Accuracy of Multiple Blood Tests to Diagnose Sepsis in Adult Burn Patients
Acronym: BioBurnSepsis
Status: Not yet recruiting | Type: Observational
Sponsor: Dohern Kym (Other)
Responsible Party: Sponsor-Investigator, Dohern Kym, Attending Physician, Burn Intensive Care Unit, Hangang Sacred Heart Hospital
Organization: Hangang Sacred Heart Hospital (Other)
Other Study IDs: 2025-020
Record Dates: First submitted 2025-08-06; First posted 2025-08-17 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Sepsis - to Reduce Mortality in the Intensive Care Unit; Burns Involving 20% or More of Body Surface
Keywords: presepsin; diagnostic accuracy; biomarker evaluation; Serum Amyloid A

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year

GROUPS / COHORTS (1):
- Burn patients with suspected sepsis: Adults ≥18 years with ≥20% TBSA burns admitted to the Burn Intensive Care Unit who developed clinically suspected sepsis (≥2 SIRS criteria)

SUMMARY:
This prospective diagnostic accuracy study evaluates the performance of presepsin and C-reactive protein (CRP) as early biomarkers for suspected sepsis in adult burn patients. From January 2021 to December 2022, 370 patients with ≥20% total body surface area burns admitted to the Burn Intensive Care Unit at Hallym University Hangang Sacred Heart Hospital were screened; 221 met inclusion criteria. At each clinical suspicion of sepsis (≥2 SIRS criteria), venous blood was drawn for simultaneous measurement of presepsin (via chemiluminescent immunoassay) and CRP (via immunoturbidimetric assay). Diagnostic accuracy will be quantified by sensitivity, specificity, positive/negative predictive values, and area under the ROC curve. The goal is to determine whether presepsin outperforms CRP for early sepsis detection in severe burn patients.

DETAILED DESCRIPTION:
Background and Rationale Sepsis is a leading cause of mortality in patients with severe burns, yet its early diagnosis is challenging. The systemic inflammatory response triggered by the burn injury itself often mimics the clinical signs of sepsis, confounding diagnosis and leading to delayed or unnecessary antibiotic use. Conventional biomarkers like C-reactive protein (CRP) and procalcitonin (PCT) lack specificity in this population, as they are elevated by the sterile inflammation from the burn itself. This study aims to overcome these limitations by evaluating the diagnostic utility of a multi-biomarker panel, analyzing their dynamic changes over time, and leveraging machine learning to develop a more accurate and interpretable diagnostic model for sepsis in burn patients.

Study Design and Objectives This is a single-center, prospective observational cohort study conducted at the Burn Intensive Care Unit (BICU) of Hallym University Hangang Sacred Heart Hospital. The study will run from September 2025 to August 2026.

Primary Objective: To evaluate the diagnostic accuracy (sensitivity, specificity, AUC) of a multi-biomarker panel-comprising Serum Amyloid A (SAA), Procalcitonin (PCT), Presepsin (PSP), and CRP-for diagnosing sepsis in adult burn patients, using the Sepsis-3 criteria as the reference standard.

Secondary Objectives: To compare the diagnostic performance of the multi-biomarker panel against individual biomarkers and standard clinical severity scores (e.g., SOFA score).

To assess the panel's ability to predict disease severity and mortality (28-day and 90-day).

To develop a predictive model for sepsis using machine learning and interpret the model's decisions using SHAP (SHapley Additive exPlanations) analysis.

Methods and Analysis Data and Sample Collection: For enrolled patients, comprehensive clinical data-including demographics, burn characteristics (%TBSA, inhalation injury), severity scores (SOFA, APACHE II), and microbiological results-will be collected. Blood samples for biomarker analysis will be collected upon ICU admission (baseline), at the time of clinical suspicion of sepsis, and serially thereafter (daily if possible) for a minimum of seven days to capture the temporal dynamics of the biomarkers.

Biomarker Panel: The core panel includes SAA, PCT, PSP, and CRP, supplemented by routine hematological markers like WBC, platelet count, NLR, and PLR.

Statistical and Advanced Analytical Plan:

Diagnostic Accuracy: Traditional statistical methods, including ROC curve analysis and DeLong's test, will be used to compare the diagnostic performance of individual and combined biomarkers.

Dynamic Analysis: To analyze the longitudinal biomarker data, generalized estimating equations (GEE) or linear mixed models (LMM) will be employed. This will allow for the quantitative assessment of biomarker trends (e.g., rate of change) and their association with sepsis diagnosis and prognosis.

Machine Learning and Interpretation: A key component of this study is the development of advanced predictive models using machine learning algorithms (e.g., Random Forest, XGBoost). To address the "black box" nature of these models, we will utilize SHAP analysis to provide transparent interpretations. This will quantify the precise contribution of each biomarker to individual patient predictions, offering deeper clinical insights into the pathophysiological state.

Sample Size: A total of 165 patients will be recruited. This sample size was calculated using G*Power software to achieve 80% power at a significance level of 0.05, assuming an expected sensitivity of 90% and specificity of 80% for the multi-biomarker panel in ROC analysis.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older.
* Admission to the Burn Intensive Care Unit (BICU) with a burn injury covering ≥10% of the Total Body Surface Area (TBSA).
* Undergoing a blood culture due to clinical suspicion of sepsis (e.g., fever, abnormal white blood cell count, hemodynamic instability) during the ICU stay.
* The participant or their legally authorized representative has provided written informed consent.

Exclusion Criteria:

* Pregnancy.
* Pre-existing immunological conditions that, in the investigator's judgment, could interfere with biomarker interpretation (e.g., long-term use of immunosuppressants, congenital immunodeficiency).
* Inability to participate at the time of study-related blood collection due to initial emergency surgery, major trauma, or significant hemorrhage.
* Any other condition for which the principal investigator deems participation to be inappropriate or unsafe for the patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults (≥18 years) with severe thermal burns (TBSA ≥20%) admitted to a single-center BICU who developed clinically suspected sepsis (≥2 SIRS criteria) during the enrollment period; all participants underwent standardized blood sampling for presepsin and CRP assays
Sampling Method: Non-Probability Sample
Enrollment: 165 (Estimated)
Dates: Start 2025-08-15 (Estimated); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy of presepsin for early sepsis detection | At the time of clinical suspicion of sepsis (Day 0), and daily for the following 7 days (Day 1 through Day 7).
  Sensitivity and specificity of presepsin (measured by chemiluminescent immunoassay on PATHFAST analyzer) for diagnosing clinically suspected sepsis (≥2 SIRS criteria) in adult burn patients.

SECONDARY OUTCOMES:
Area under the ROC curve (AUC) for presepsin versus CRP | Through study completion, an average of 1.5 years.
  Comparison of AUCs for presepsin and CRP using DeLong's test to assess which biomarker better discriminates sepsis versus non-sepsis.